CLINICAL TRIAL: NCT01563926
Title: An Open, Multi-Centre Trial Evaluating Acceptance of the New Liquid Growth Hormone Formulation - Norditropin Simplexx™ in Children With GH Deficiency
Brief Title: Evaluating Acceptance of New Liquid Somatropin Formulation in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1315
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Genetic Disorder; Turner Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Dosed by individual needs as judged by the Investigator (trial physician). Injected subcutaneously (s.c./under the skin)

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to evaluate the new liquid somatropin formulation in children with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent by patient and/or guardian/parents
* Patients with one of the following diagnosis: Growth failure due to growth hormone deficiency (GHD), Turner syndrome, or growth retardation in children with chronic renal disorders
* Patients who are willing to inject themselves and answer questionnaires or young patients whose parents/guardian are willing to inject their child and answer questionnaires
* Patients on growth hormone therapy for at least 6 weeks before entering the trial

Exclusion Criteria:

* Pregnancy or breast feeding women
* Suspected or known allergy to trial product
* Other daily injection therapy (non-growth hormone, e.g insulin-therapy)
* Participating in any other trial involving other investigational products within the last 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2000-10-23 (Actual); Primary Completion 2002-10-10 (Actual); Study Completion 2002-10-10 (Actual)

PRIMARY OUTCOMES:
Patient acceptance of the new liquid growth hormone formulation

SECONDARY OUTCOMES:
Number of Adverse Events (AE)
Number of Serious Adverse Events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Israel (6):
  - Novo Nordisk Investigational Site, Afula
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
  - Novo Nordisk Investigational Site, Tel Aviv

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com